CLINICAL TRIAL: NCT03749590
Title: Prospective Randomized Controlled Phase III Trial to Investigate the Efficacy of Magnesium Sulfate in the Prevention of Post-ERCP Pancreatitis.
Brief Title: Magnesium Sulfate in the Prevention of Post-ERCP Pancreatitis.
Acronym: MagPEP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The design of the MagPEP trial is no longer in compliance with the current state of science.
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MagPEP; 2009-013294-18 (EudraCT Number)
Record Dates: First submitted 2018-11-12; First posted 2018-11-21 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Post-ERCP Pancreatitis
Keywords: MagPEP, post-ERCP pancreatitis, Magnesium Sulfate
MeSH Terms: interventions — Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Magnesium (Experimental): Patients receive 2 infusions of 500 ml NaCl 0,9%: the first one 60 min before ERCP and the second one 6 hours after ERCP.
  With each infusion 10 ml magnesium sulfate (4930 mg magnesium sulfate = 20 mmol magnesium) are administered (total dose: 9860 mg magnesium sulfate).
  Interventions: Drug: Magnesium Sulfate
- Placebo (NaCl 0,9%) (Placebo Comparator): Patients receive 2 infusions of 500 ml NaCl 0,9%: the first one 60 min before ERCP and the second one 6 hours after ERCP.
  To each infusion 10 ml NaCl 0.9% (Placebo) will be added .
  Interventions: Drug: Placebo (NaCl 0,9%)

INTERVENTIONS:
Drug: Magnesium Sulfate — Patients receive 2 infusions (10 ml magnesium sulfate added to 500 ml NaCl 0.9%): the first infusion 60 min before and the second one 6 hours after ERCP
  Other Names: Magnesium Sulfate Heptahydrate
  Arms: Magnesium
Drug: Placebo (NaCl 0,9%) — Patients receive 2 infusions (10 ml NaCl 0.9% added to 500 ml NaCl 0.9%): the first infusion 60 min before and the second one 6 hours after ERCP
  Arms: Placebo (NaCl 0,9%)

SUMMARY:
MagPEP is a multi-centre, randomized, phase III, double blind, placebo controlled, parallel group trial. It evaluates magnesium sulfate for the prevention of post-ERCP pancreatitis. Adult patients with a medical indication for ERCP are to be randomized (1:1 ratio) to receive either magnesium sulfate or placebo (NaCl 0,9%) 60 min before and 6 hours after ERCP.

DETAILED DESCRIPTION:
Title: prospective, randomized, placebo controlled, phase III trial to evaluate the efficacy of magnesium sulfate for the prevention of post-ERCP pancreatitis

Study drug: Magnesium sulfate

Indication: post-ERCP pancreatitis

Study design: multi-centre, randomized, phase III, double blind, placebo controlled, parallel group

Patient population: adult patients with a medical indication for ERCP

Number of patients: 1376 randomized to two equal groups

Treatment: patients receive 2 infusions of 500 ml NaCl 0,9%: the first one 60 min before ERCP and the second one 6 hours after ERCP. To the infusions 10 ml of either magnesium sulfate or placebo (NaCl 0,9%) will be added.

ELIGIBILITY:
Inclusion Criteria:

* medical indication for ERCP
* first ERCP in the Patient
* signed informed consent forms for ERCP and MagPEP trial

Exclusion Criteria:

* privious ERCP
* hypersensitivity to study medication or similar substances
* participation in another clinical trial during the last 4 weeks
* addictive disorders
* women who are pregnant or breastfeeding
* unwillingness or inability to comply with study protocol
* acute pancreatitis
* renal insufficiency of stage 4 or higher
* active hyperthyreosis
* symptomatic bradycardia (<35/min)
* known history of Myasthenia gravis
* AV bock > first degree or other bradycardic disorders of conductivity
* liver cirrhosis Child C
* coagulation disorder
* urinary stone diathesis (calcium magnesium ammonium phosphate stones)
* patients who are not able to provide informed consent
* intake of magnesium during the last 14 days
* intake of calcium antagonists

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2020-07 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
reduction in the incidence of post-ERCP pancreatitis by 50 % | 24 hours after ERCP

SECONDARY OUTCOMES:
reduction in intake of analgesics | during the first 24 hours after ERCP and, if a post-ERCP pancreatitis occurs, until discharge from hospital
duration of stay in hospital after ERCP | from end of ERCP to discharge from hospital; assessed on day 30 after ERCP
reduction in premature protease activation | during treatment period, assessed 24 h after ERCP
reduction in severity of post-ERCP pancreatitis | from 24 hours after ERCP onwards, assessed on day 30 after ERCP
reduction in 30-day morbidity | 30 days after ERCP

CONTACTS AND LOCATIONS:
Locations (1):
- Klinik für Innere Medizin A, Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany